CLINICAL TRIAL: NCT03155763
Title: Impact of Acute and Chronic Individual Histological Lesions and Composite Scores in Implantation Biopsies on Short-term and Long-term Kidney Allograft Outcomes
Brief Title: Histology of Implantation Biopsies and Kidney Allograft Outcomes
Acronym: KALIMBO
Status: Completed | Type: Observational
Sponsor: Andriy Trailin (Other)
Responsible Party: Sponsor-Investigator, Andriy Trailin, Head of Laboratory Diagnostics and General Pathology Department, State Institution, Zaporizhzhia Medical Academy of Post-Graduate Education Ministry of Health of Ukraine
Organization: State Institution, Zaporizhzhia Medical Academy of Post-Graduate Education Ministry of Health of Ukraine (Other)
Other Study IDs: 0105U007599
Record Dates: First submitted 2017-05-13; First posted 2017-05-16 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Kidney Graft Dysfunction
Keywords: kidney transplantation; implantation biopsy; histology; allograft function; allograft survival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Formalin-fixed paraplast-embedded kidney biopsies were retained in a biorepository.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Intraoperative kidney allograft preimplantation biopsy; Intraoperative kidney allograft postreperfusion biopsy

SUMMARY:
The morphology of transplanted kidney is considered to be important for graft outcomes in early and late posttransplant period. Individual histological lesions at the time of kidney transplantation, such as sclerosis of glomeruli, vascular narrowing and interstitial fibrosis, and composite histological lesions, which integrate histopathological findings in different compartments, showed association with suboptimal graft outcomes. However there are no consistent association between individual or composite lesions and transplant outcomes. Some possible explanations for such inconsistent results are non-uniformity in grading histological lesions or in defining graft outcomes. Furthermore, studies vary in terms of patient selection, and some results are not corrected for covariates. It is also unclear, whether acute biopsy features associated with the donor kidney can provide prognostic information, in addition to the chronic lesions? This single-center study aimed to evaluate which acute and chronic histological lesions and composite histological scores in donor kidney intraoperative biopsies alone or in combination with clinical variables are best associated with short- and long-term kidney graft outcomes, such as impairment of early kidney allograft function, immunological acute kidney allograft rejection, pyelonephritis, allograft function at 1, 3, 6, 12 months, 2, 3, 4 and 5 years, and graft survival at 1 and 5 years.

DETAILED DESCRIPTION:
130 consecutive patients with end-stage renal disease (ESRD), receiving a kidney only transplant from April 2005 to December 2010 in a single center, and having both intraoperative biopsies with ≥ 7 glomeruli and ≥ 1 arteries and complete follow-up data up to 5 years were included in the study.

Intraoperative biopsy consisted of preimplant biopsy (at the backtable, 1 core) and 30-minutes postreperfusion biopsy (1 core), which were taken in order to study the impact of ischemia/reperfusion injury on transplant outcomes and to serve a reference for subsequent biopsies.

Donor population included live donors (32.6%), ideal deceased donors (50%), expanded-criteria donors (7.9%) and 9.0% of non-heart-beating donors. Donors were subjected to donor evaluation protocol in accordance with local guidelines, including a standard clinical, instrumental and laboratory examination.

All recipients and donors were Caucasians.

Histological scoring Needle (14-18-gauge) biopsies were obtained and tissue was fixed in 10% buffered formalin and embedded in paraffin. A 3-4 µm sections of preimplant and postreperfusion kidney allograft implantation biopsies (KALIMBO) were stained for light microscopy with hematoxylin-eosin (3 slides), periodic acid-Schiff (3 slides), and Masson's trichrome (1 slide). A minimum of 21 tissue sections were examined for each biopsy. Banff-1997 criteria for posttransplant biopsies, Banff-2016 criteria for preimplant biopsies, as well as criteria suggested by Remuzzi et al. (1999) and Cosyns et al. (1998) were applied for scoring.

Based on the estimation of individual acute and chronic lesions, the acute, chronic and total posttransplant and preimplant Banff scores, Remuzzi score, and acute, chronic and total lesion indexes by Cosyns were calculated. In addition, previously published composite histological scores, such as chronic allograft damage index (CADI), donor damage score (DDS), chronic damage score (CDS), and interstitial fibrosis and fibrous thickening score (CIV) were computed.

Clinical risk factors and outcomes examined The analysis was performed 60 months later after the last transplant in the study population. Donor, graft and recipient characteristics and transplant outcomes were extracted from archival patient records and outpatient cards blinded to all pathologic data. Data were retrieved on donor source, sex and age, and cause of death, donation after cardiac death or expanded criteria donation for deceased donors.

Recipient's pretransplant variables included: age, gender, cause of ESRD, body mass index (BMI), dialysis modality and duration, previous transplants, and presence of chronic arterial hypertension, defined as a regular intake of antihypertensive drugs. The information related to transplantation (cold ischemia time and second warm ischemia time) was also obtained. Posttransplant data retrieved were limited to initial graft function (immediate, delayed or slow), and the number and time of occurrence of acute rejection episodes or pyelonephritis, and time of graft failure defined as return to dialysis therapy.

All recipients received triple maintenance immunosuppressive therapy consisting of calcineurin-inhibitor (cyclosporine or tacrolimus), mycophenolate mofetil, and steroid. Each patient, enrolled in this study, was followed for five years until death/return to dialysis or until December 2015.

The end points of the study were impairment of early kidney allograft function, immunological acute kidney allograft rejection, pyelonephritis, allograft function at 1, 3, 6, 12 months, 2, 3, 4 and 5 years, and graft survival at 1 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* adult kidney transplant recipients who underwent transplantation at Zaporizhzhia Transplant Center;
* cadaveric or living single kidney only transplant;
* informed written consent;
* adequate intraoperative biopsy (in total ≥ 7 glomeruli and ≥ 1 arteries in preimplant and postreperfusion biopsies);
* complete follow-up data up to 5 years.

Exclusion Criteria:

* not consent with research;
* non-complete follow-up data up to 5 years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All recipients and donors were Caucasians and Ukrainians.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2005-04-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Five-year death-censored kidney allograft survival | Five years
  The time of graft failure was defined as return to dialysis therapy

SECONDARY OUTCOMES:
Delayed graft function | The day 8
  Delayed graft function was defined as the need for dialysis in the first postoperative week without evidence of acute rejection or pyelonephritis
Slow graft function | The day 8
  Slow graft function was defined as serum creatinine on day seven ≥300 μmol/L without evidence of acute rejection or pyelonephritis.
Acute rejection | During five years
  Acute rejection was defined by characteristic clinical symptoms and ultrasound findings and by the need for treatment, with or without biopsy confirmation.
Pyelonephritis | During five years
  Pyelonephritis was defined by characteristic symptoms, a urine sediment analysis, and a urinary culture test.
Allograft function at 1, 3, 6, 12 months, 2, 3, 4 and 5 years | During five years
  Allograft function at 1, 3, 6, 12 months, 2, 3, 4 and 5 years was assessed with glomerular filtration rate (CKD-EP equation).
One-year death-censored kidney allograft survival | One year
  The time of graft failure was defined as return to dialysis therapy

CONTACTS AND LOCATIONS:
Overall Officials: Andriy V Trailin, MD, DSc, Principal Investigator — State Institution, Zaporizhzhia Medical Academy of Post-Graduate Education Ministry of Health of Ukraine
Locations (1):
- Laboratory Diagnostics and General Pathology Department, State Institution "Zaporizhzhia Medical Academy of Post-Graduate Education Ministry of Health of Ukraine", Zaporizhzhia, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
We are going to share raw data on kidney baseline histology, graft function and survival up to 5 years after the publication of all results obtained. IPD will be available through an open access repository of data (ClinicalTrials.gov)